CLINICAL TRIAL: NCT04692207
Title: Prostate Biopsies With Target Lesion on MRI : When Can Non-targeted Biopsies be Dispensed With
Brief Title: Prostate Biopsies With Target Lesion on MRI
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0684
Record Dates: First submitted 2020-12-28; First posted 2020-12-31 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Prostate Cancer
Keywords: Targeted prostate biopsy; Non-targeted prostate biopsy; MRI; prostate; biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our objective is to search for clinical, biological and imaging element that would better define the patient population that could benefit from targeted prostate biopsies only (from a cohort of patients who had targeted and non-targeted prostate biopsies).

ELIGIBILITY:
Inclusion criteria:

* Age > or = at 18 years old
* Prostatic MRI performed at the Montpellier University Hospital
* Realization of targeted prostate biopsies (by fusion of MRI - ultrasound images) and non-targeted biopsies

Exclusion criteria:

* Pre-biopsy MRI performed outside of the Montpellier University Hospital
* MRI with artefacts
* Not performing 12 non-targeted prostate biopsies

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had a prostate MRI between June 2017 and March 2020 for suspected cancer, followed by targeted and non-targeted prostate biopsies (12) at the Montpellier University Hospital
Sampling Method: Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Non-targeted biopsy not finding cancer of finding cancer of a grade lower than or egal to that found on targeted biopsies | 1 month
  Non-targeted biopsy not finding cancer of finding cancer of a grade lower than or egal to that found on targeted biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Millet, PUPH, Study Director — University Hospital, Montpellier
Locations (1):
- University hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC